CLINICAL TRIAL: NCT06396416
Title: Obesity Management for Kidney TRANSPLANTation: a Vanguard Study for an Innovative Randomized Controlled Trial, Embedded in Routine Care (OK-TRANSPLANT 2)
Brief Title: Obesity Management for Kidney TRANSPLANTation: OK-TRANSPLANT 2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Queen Elizabeth II Health Sciences Centre (Other); St. Michael's Hospital (Toronto, Canada) (Unknown)
Responsible Party: Principal Investigator, Kristin Clemens, Associate Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OK-TRANSPLANT 2
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Chronic Kidney Disease
Keywords: Weight Management; Transplant; GLP-1RA; Pilot Study; Registries; Pragmatic
MeSH Terms: conditions — Obesity; Renal Insufficiency, Chronic | interventions — semaglutide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Weight Management Program (Experimental): A maximum tolerated dose of semaglutide (Ozempic/Wegovy) will be administered once weekly subcutaneously, up to a dose of 2.0 mg. Participants will also receive nutritional and movement advice, as well as virtual coaching once every 4 weeks for 6 months.
  Interventions: Drug: Semaglutide; Behavioral: Virtual Weight Management Coaching
- Usual Care (No Intervention): Usual care participants will continue to receive the typical standard of kidney and diabetes care. They will not receive any study medication or coaching.

INTERVENTIONS:
Drug: Semaglutide — Maximum tolerated dose of semaglutide subcutaneously once weekly. Maximum dose of 2.0 mg.
  Other Names: GLP-1RA; Ozempic; Wegovy
  Arms: Virtual Weight Management Program
Behavioral: Virtual Weight Management Coaching — Virtual meeting with intervention coach once every 4 weeks for 6 months, where the coach will discuss the goals and progress with participant, nutritional advice, exercise advice, and motivational support.
  Arms: Virtual Weight Management Program

SUMMARY:
OK-TRANSPLANT 2 is a vanguard study for a large randomized, pragmatic, open-label trial.

We will randomize participants with obesity, high-risk CKD/dialysis who are hoping for lose weight for the purpose of kidney transplant. Subjects will either be enrolled on a virtual weight management program or continue their usual care.

DETAILED DESCRIPTION:
Obesity is well-recognized as an independent risk factor for chronic kidney disease (CKD) including end-staged kidney disease (ESKD). In people with ESKD, obesity can preclude access to lifesaving kidney transplantation. Of solid organ transplant programs in Canada, 80% exclude people with obesity (based upon body mass index or BMI), due to a potential risk of perioperative complications and post-transplant mortality.

Losing weight for kidney transplantation can, however, be extremely difficult. Medications that can promote weight loss in other populations including glucagon-like peptide 1 receptor agonists (GLP-1RA; liraglutide, semaglutide, and dulaglutide) and glucose-dependent insulinotropic polypeptide (GIP-1RA)/GLP-1RAs (tirzepatide), have not been studied in devoted trials of advanced CKD participants, and their efficacy and safety remain unclear.

Nutritional advice is often very difficult to follow when trying to balance kidney and diabetes diets (e.g. potassium), and if diets are too restrictive, there may be protein-energy wasting which could be detrimental to patients. People with high-risk CKD frequently live with functional impairment which can limit exercise. Weight loss programs can be cost prohibitive to those who are already socioeconomically disadvantaged.

A vanguard is needed before a large, multicentered RCT: A feasibility study will allow us to ensure that we can recruit a sufficient sample of participants into our trial, that our trial processes are inclusive, and that they are acceptable to patients. In the vanguard phase of our trial, we will answer the following questions:

1. Is participant recruitment into a large multi-centered trial feasible?
2. Will participants remain adherent to their assigned treatment arm over 26 weeks of study?
3. Will participants find our program acceptable?
4. Will safety events preclude us from testing our intervention in a larger RCT?

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* BMI > 35 kg/m^2
* >10% risk of ESKD requiring renal replacement therapy over 2 years or receiving dialysis

Exclusion Criteria:

* Known contraindication to a GLP-1RA
* Type 1 diabetes
* No access to semaglutide via drug coverage
* Absolute contraindication to kidney transplant
* Pregnant, breastfeeding or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 12 months
  Number participants recruited within 12 months of trial initiation at each centre

SECONDARY OUTCOMES:
Adherence to Scheduled Coaching Visits | 26 weeks
  Percentage of participants randomized to the intervention attend >75% of their scheduled coaching visits.
Adherence to Study Medication | 26 weeks
  Percentage of participants randomized to the intervention fill >75% of their semaglutide prescriptions.
Crossover of Intervention and Control | 26 weeks
  Percentage of participants randomized to the usual care group who are started on a GLP-1RA medication or other weight loss intervention during the study
Adverse events | 26 weeks
  Percentage of participants that experience acute kidney injury (AKI), hypoglycemia, gastrointestinal side effects.

OTHER OUTCOMES:
Percentage of Change in HbA1c | 26 weeks
  Percentage of change in HbA1c from baseline to 26 weeks
Change in 2-week mean fasting glucose | 26 weeks
  Change in 2-week mean fasting glucose (mmol/L) from baseline to 26 weeks
Change in 2-week glycemic variability and time in range (TIR) | 26 weeks
  For those using a Libre or Continuous Glucose Monitoring at baseline, Percentage of change in 2-week glycemic variability and time in range from baseline to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristin K Clemens, MD, MSc, Principal Investigator — St. Joseph's Health Care London; Louise Moist, MD, MSc, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No